CLINICAL TRIAL: NCT02417402
Title: Efficacy of Educating Physical Therapists on Clinical Practice Guidelines and Pain Management in the Treatment of Patients With Nonspecific Chronic Low Back Pain: a Cluster Randomized Controlled Trial
Brief Title: Efficacy of Educating Physical Therapists in the Treatment of Patients With Nonspecific Chronic Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We had many issues related to recruitment. After many attempts we want to suspend the study with 13 patients.
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo Rossi Nogueira Rizzo, Masters student, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNICID032015
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Back Pain
Keywords: back pain; low back pain; chronic low back pain
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Trained Immunity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Untrained Physical Therapists (Active Comparator): The patients allocated to the Control group will be treated by physical therapists who did not receive any training about clinical practice guidelines and pain management. These patients will receive the usual care from their physical therapists.
  Interventions: Other: Control
- Trained Physical Therapists (Experimental): The patients allocated to the Experimental group will be treated by physical therapists who received training about clinical practice guidelines and pain management.
  Interventions: Other: Trained

INTERVENTIONS:
Other: Control — The patients allocated to the Control group will be treated by physical therapists who did not carry out the training before treatment. The physical therapists will use their usual care for nonspecific chronic low back pain. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week). Each treatment session has an estimated duration of 50-60 minutes.
  Other Names: physical therapist education; guidelines implementation
  Arms: Untrained Physical Therapists
Other: Trained — The patients allocated to the Experimental group will be treated by physical therapists who carried out the training before treatment. The training will be designed to guide the physical therapists beliefs and attitudes to a biopsychosocial model; update knowledge contained in clinical practice guidelines; and enable physical therapists to identify, integrate and address psychosocial factors in patients with nonspecific chronic low back pain. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week). Each treatment session has an estimated duration of 50-60 minutes.
  Other Names: physical therapist education; guidelines implementation
  Arms: Trained Physical Therapists

SUMMARY:
The aim of this trial is to investigate if patients treated by physical therapists who received an update on clinical practice guidelines and pain management have better outcomes than patients treated by physical therapists who did not received such training.

DETAILED DESCRIPTION:
The training "Update on the treatment of patients with nonspecific chronic low back pain" will be announced in the social network by members of the study. Interested physical therapists will send an email to one of the study authors with their information regarding the inclusion criteria. After two months of notice, interested and eligible physiotherapists will be randomized into two groups of 15 participants each.

The study arms are: 1) control group (physical therapist who will not receive training) and 2) experimental group (physical therapist who will receive training). Before and after training, attitudes, beliefs and knowledge about low back pain guidelines will be evaluated.

Each physical therapist will recruit for the study a total of fifteen consecutive patients with chronic nonspecific low back pain (total sample=150 patients). All the patients will be assessed before the first session by a blinded examiner who will be unaware about the group allocation.

Clinical outcomes (pain, disability, fear avoidance beliefs and pain catastrophizing) will be collected at baseline and at 5 weeks, 3 and 6 months after randomization. All statistical analysis will be conducted following the principles of intention to treat analysis and the between-group differences will be performed using Mixed Linear Models.

ELIGIBILITY:
Inclusion Criteria:

* patients seeking care for chronic non-specific low back pain (defined as pain or discomfort between the costal margins and the inferior gluteal folds, with or without referred symptoms in the lower limbs, for at least 3 months), with a pain intensity of at least 3 points measured by a 0-10 pain numerical rating scale, aged between 18 and 65 years.
* physiotherapists who treat exclusively patients with musculoskeletal pain, duly accredited by the National Council of Physical Therapy, physiotherapists offering private or medical insurance treatment individually to their patients, lasting 50-60 minutes each session, physiotherapists from 2 to five years of graduation and / or working in the area for the same period, that treat at least 2 patients with low back pain per month, and who are willing to treat at least 10 patients for the study.

Exclusion Criteria:

* patients will be excluded if they have any contraindication to physical exercise or ultrasound or short wave therapy, evidence of nerve root compromise (i.e one or more of motor, reflex or sensation deficit), serious spinal pathology (such as fracture, tumor, inflammatory and infectious diseases), serious cardiovascular and metabolic diseases, previous back surgery and pregnancy.
* physiotherapists who want to stop the activities for some reason that prevents participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Pain NRS) | 5 weeks after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability (24-item Roland Morris Disability Questionnaire) | 5 weeks after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain intensity (Pain NRS) | 3 and 6 months after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability ( 24-item Roland Morris Disability Questionnaire) | 3 and 6 months after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire
Fear Avoidance Beliefs (FABQ) | 5 weeks, 3 months and 6 months after randomization
  Fear avoidance belief will be measured by the 16-item Fear Avoidance Belief Questionnaire (FABQ)
Pain Catastrophizing (PCS) | 5 weeks, 3 months and 6 months after randomization
  Pain Catastrophizing will be measured by the 13-item Pain Catastrophizing Scale (PCS)

OTHER OUTCOMES:
Pain attitudes and beliefs for physiotherapists (PABS.PT) | Baseline and 5 weeks after randomization
  Pain Attitudes and Beliefs will be measured by the 19-item Pain Attitudes and Beliefs Scale for Physiotherapists (PABS.PT)
Adherence to guidelines for physiotherapists (0-100% Low Back Pain Vignettes) | Baseline and 5 weeks after randomization
  Adherence to guidelines for physiotherapist will be measured by the 0-100% Low Back Pain Vignettes

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo OP Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo